CLINICAL TRIAL: NCT05470179
Title: Changes in Arch Parameters After Molar Distalization; Hybrid Hyrax Distalizer Versus Pendulum in Adolescent Class II Patients Prospective Randomized Clinical Study
Brief Title: Changes in Arch Parameters After Molar Distalization; Hybrid Hyrax Distalizer Versus Pendulum
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Abdelrhman Shendy Abdelrhman (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdelrhman Shendy Abdelrhman, Lecturer, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 824/220
Record Dates: First submitted 2022-07-04; First posted 2022-07-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Angle Class 2 Malocclusion
Keywords: hybrid hyrax distalizer; Pendulum distalizer; class II division 1 and 2; molar distalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid hyrax distalizer (Active Comparator): Inverted hyrax with 2 miniscrews for 6 months for maxillary molar distal movement in class II angle malocclusion
  Interventions: Device: Hybrid hyrax distalizer; Device: Pendulum distalizer
- Pendulum distalizer device (Active Comparator): Modified pendulum with miniscrews for 6 months for maxillary molar distal movement in class II angle malocclusion
  Interventions: Device: Hybrid hyrax distalizer; Device: Pendulum distalizer

INTERVENTIONS:
Device: Hybrid hyrax distalizer — class 2 Angle malocclusion
Device: Pendulum distalizer — class 2 Angle malocclusion

SUMMARY:
this study was to compare the changes in arch parameters after molar distalization; hybrid hyrax distalizer versus Pendulum distalizer using CBCT.

DETAILED DESCRIPTION:
Evaluation of maxillary molar amount of distal movement and the amount of anchorage loss Arch length, arch width, arch depth

ELIGIBILITY:
Inclusion Criteria:

* For group 1(Hybrid hyrax distalizer) Patients suffering maxillary collapse with a skeletal background with unilateral or bilateral posterior crossbite.
* For group 2 (Pendulum distalizer) Patients with skeletal class I or class II malocclusion who needed upper first and second molar distalization for incisor retraction or relieving of the upper arch crowding and minimum or no crowding in lower jaw were selected.
* All Patients had no systemic diseases that may affect bone quality or interfere with orthodontic treatment, periodontal disease and no previous orthodontic treatment.
* Age range was 13 to 17 years.

Exclusion Criteria:

* Missed upper first molar.
* un-cooperative patient

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Angles in degree SNA,SNB,ANB, Molar Rotation | 6 months
  Using cbct and cast
Arch parameters in millimeter Arch length, width,depth and circumference | 6 Months
  Assessment of airway using cbct

SECONDARY OUTCOMES:
Nasopharyngeal airway dimensions in Cubic centimeters | 6 months
  CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AE Shendy, Principal Investigator — Lecturer - Orthodontic department -faculty of dental medicine -Al-Azhar university
Locations (2):
- Egypt (2):
  - Mohamed Shendy, Cairo, Nasr City
  - Cairo, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Comparison between two techniques of molar distalization
Supporting Information: Study Protocol, ICF
Time Frame: 6 Months
Access Criteria: shendy_ortho@azhar.edu.eg

REFERENCES:
- [Background] Bishara SE, Staley RN. Maxillary expansion: clinical implications. Am J Orthod Dentofacial Orthop. 1987 Jan;91(1):3-14. doi: 10.1016/0889-5406(87)90202-2. PMID 3541577
- [Background] Haas AJ. Palatal expansion: just the beginning of dentofacial orthopedics. Am J Orthod. 1970 Mar;57(3):219-55. doi: 10.1016/0002-9416(70)90241-1. No abstract available. PMID 5263785